CLINICAL TRIAL: NCT01779960
Title: Understanding in Depth the Physical Inactivity of Patients With COPD: Comparison of the Summer-Winter Variability in the Level of Physical Activity in Daily Life in Brazilian and Belgian Patients
Brief Title: Summer-Winter Variability in the Level of Physical Activity in Daily Life in Brazilian and Belgian Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Fabio Pitta, PhD, Fabio Pitta, Universidade Estadual de Londrina
Other Study IDs: LFIP-001-KCF-1; 483107/2011-5 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Motor activity; Climatologic station
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Londrina: 20 patients with moderate-severe COPD from State University of Londrina, Brazi
  Interventions: Other: Londrina
- Leuven: 20 patients with moderate-severe COPD from Catholic University of Leuven, Belgium
  Interventions: Other: Leuven

INTERVENTIONS:
Other: Londrina — Two groups of patients, one group in Londrina and another group in Leuven, will be simultaneously and objectively evaluated concerning their physical activity in daily life during one week in two different moments: in January 2013 (winter in Leuven and summer in Londrina), and then the same two groups of patients will be once again simultaneously re-evaluated during another week in July 2013 (summer in Leuven and winter in Londrina).
  Other Names: Climatologic Station
  Groups: Londrina
Other: Leuven — Two groups of patients, one group in Londrina and another group in Leuven, will be simultaneously and objectively evaluated concerning their physical activity in daily life during one week in two different moments: in January 2013 (winter in Leuven and summer in Londrina), and then the same two groups of patients will be once again simultaneously re-evaluated during another week in July 2013 (summer in Leuven and winter in Londrina).
  Other Names: Climatologic Station
  Groups: Leuven

SUMMARY:
Up to this moment, the majority of studies assessing the level of physical activity in daily life in patients with COPD are limited to a cross-sectional design, which does not take into account natural variation of physical activity in daily life due to differences in climatic conditions faced throughout the year. Preliminary evidences suggest that patients with COPD have different physical activity levels according to the seasons of the year. However, the limited current evidences do not allow us to know the magnitude of differences in the level of daily physical activity in patients with COPD when taking into account climatic changes resulting from different seasons of the year in cities and countries with contrasting climatic conditions. This gap observed in the literature does not allow us at this moment to know whether we should or not consider the season of the year as one of the main causes of variability while assessing physical activity in daily life in patients with COPD.

The present project proposes to investigate the hypothesis that patients with COPD who live in a place with less marked decrease in temperature between summer and winter (Londrina, Brazil) have less variability in the level of physical activity in daily life through the year in comparison to patients who live in a place with more marked climatic variability during these seasons (Leuven, Belgium).

DETAILED DESCRIPTION:
The sample will be composed by at least 20 patients with moderate-severe COPD from each institution involved (Catholic University of Leuven, Belgium and State University of Londrina, Brazil), adding up to 40 patients (see sample size calculation below). However, the sample size could be increased if necessary to achieve intermediate calculation of the sample power performed during the study. Both groups should be similar concerning anthropometric characteristics, gender distribution and severity feature of the disease (especially FEV1). Therefore, an eventual increase in the final number of patients may also be necessary in case this similarity is not achieved in the final data collection of the planned sample.

Data collection will be performed in the Laboratory of Research in Respiratory Physiotherapy from the State University of Londrina (Londrina, Brazil) and in the University Hospital Gasthuisberg from the Catholic University of Leuven (Leuven, Belgium).

The study has a longitudinal design. Two groups of patients, one group in Londrina and another group in Leuven, will be simultaneously and objectively evaluated concerning their physical activity in daily life during one week in two different moments: in January 2013 (winter in Leuven and summer in Londrina), and then the same two groups of patients will be once again simultaneously re-evaluated during another week in July 2013 (summer in Leuven and winter in Londrina). Changes in the level of physical activity in daily life between summer and winter in the two groups will then be compared. Monitoring of physical activity in daily life: two activity monitors (the SenseWear armband and the Fitbit) will be simultaneously worn during 7 consecutive days. The SenseWear armband (BodyMedia, Pittsburg, PA, USA) is a multisensor composed by a biaxial accelerometer and physiologic sensors. It is a small (8.8 x 5.6 x 2 cm) and lightweight (82g) monitor that is worn at the upper right arm and was already validated for energy expenditure estimation in patients with COPD [12,13]. The Fitbit (Fitbit, Inc., San Francisco, CA, USA) is a recently released triaxial accelerometer that is smaller (3.6 x 2.9 x 1 cm) and more lightweight (8g) than the SenseWear. According to the manufacturer, the Fitbit can be used in different positions, including at the waist. This device provides the number of steps, the distance walked and the energy expenditure in calories, among other variables. In the 7 days of assessment, the patient will remain with the device during 24 hours/day. The patients will be strictly instructed to avoid changing their daily physical activity habits during the monitoring period.

To characterize the sample, all patients will be submitted to spirometry, 6 minute walking test (6MWT) and quality of life assessment (Chronic Respiratory Disease Questionnaire - CRQ), also described in detail in the subsection "Methods".

For each patient, further information will be also registered: types of drugs used by the patient, their dosage and how often these drugs are used in the last month before inclusion in the study; characterization of the history of acute exacerbations occurred in the last year (if it is the case); presence of respiratory insufficiency on admission or during the study period (PaO2 < 60 mmHg and/or SpO2 < 90% with or without PaCo2 > 50 mmHg, breathing on room air); need for long-term oxygen supplementation previously or during the study period; practice or not of regular physical activity in the last year.

LOGISTICS INVOLVED IN DATA COLECTION IN BOTH CENTERS

In the first period of data collection (January 2013), the Brazilian coordinator of the project (Prof. Fabio Pitta) will travel to Leuven to participate in data collection and organization on site. The Brazilian project coordinator will arrive in Leuven two weeks before the data collection, and in conjunction with the Belgian coordinator of the project (Prof. Thierry Troosters) and the European researchers will prepare all necessary logistic actions to ensure the adequate performance of the study. After the preparation period, data collection itself will be performed in three weeks, with 15 patients being assessed in the first week and 14 in the third week. Spirometry, 6MWT and CRQ will be performed on Friday, and data collection of physical activity will be performed from Saturday to next week's Saturday. The 1-week interval between the first and second weeks of assessment will be used to download the data and discuss eventual issues raised in the first week of assessment, and thus this justifies the need of 15 activity monitor devices (SenseWear and Fitbit) in each center adding up to 60 necessary devices (as data collection will simultaneously occur in both centers).

Previously, the Brazilian team involved in the project will be prepared by the Brazilian coordinator with the same instruction, since the first period of data collection in Londrina will occur simultaneously with Leuven. Therefore, the first period of data collection in Londrina will be performed by the Brazilian researchers involved in the study, coordinated from Leuven by Prof. Fabio Pitta. The research team will make sure that the Brazilian researchers are prepared and trained to perform all assessments, including the objective quantification of physical activity in daily life, as well as the identical application of the 6MWT and CRQ in both centers.

In the second phase of data collection (July 2013), the European and the Brazilian researchers will be responsible for the assessments with the same protocol trained and performed in the first phase of data collection. Therefore, Prof. Fabio Pitta will coordinate the data collection in Londrina while Prof. Thierry Troosters will coordinate the data collection in Leuven to ensure the reproducibility of all the methods in the second data collection moment..

After the second phase of data collection, further project activities will have the coordination centralized in Londrina, with the Brazilian coordinator of the project.

STATISTICAL ANALYSIS AND SAMPLE SIZE CALCULATION

Statistical analysis will be performed using the SPSS v. 17 Statistical Package (SPSS, Inc., Chicago IL, EUA) and the GraphPad Prism 5.0 (GraphPad Software Inc., San Diego, CA, EUA). The Shapiro-Wilk test will be initially used to analyze the normality in data distribution. In case of variables normally distributed, data will be described as mean ± standard deviation, and those variables with non-normal distribution will be described as median [25%-75% interquartile range]. Summer-winter changes in the same group of patients will be analyzed by the paired t test (parametric analysis) or the Wilcoxon test (non-parametric analysis). Summer-winter differences between the two groups of patients (Londrina and Leuven) will be analyzed by the unpaired t test (parametric analysis) or by the Mann-Whitney (non-parametric analysis). Variables of spirometry, 6MWT and CRQ of both groups will be analyzed by the unpaired t test in the two assessment moments. Correlations will be analyzed by the Pearson or Spearman coefficient, depending on the normality on data distribution. For all analysis, statistical significance will be set at p less than 0.05.

The sample size of the study was calculated according to the assumption of a mean (and standard deviation) difference of counts/day between two groups of patients with COPD, being one in Europe and one in Brazil. The first group was assessed in the summer and winter, as found in the study by Sewell et al. performed in England [10]. This study presented a mean difference of 5656 counts (8857 in summer and 3201 in winter), with a standard deviation of 7497 and 2629 counts, respectively. The second group was based on our hypothesis that there will be no (or little) change in physical activity in daily life due to seasonal variation in Londrina (Brasil) based on the study by Probst et al. (Respiratory Care 2011; 56[11]: 1799-87), taking into account a similar standard deviation of 5063 counts/day. With a power of 90%, alfa coefficient of 0.05, at least 12 patients in each group will be necessary to detect significant difference in the level of physical activity in daily life between summer and winter within the groups. Taking into account an eventual difficult setting with drop-out rate of 40% due to difficulties in the data collection protocol involving the motion sensors, a minimum of 20 patients will be included to compose either group (Londrina and Leuven), adding up to 40 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD based on internationally accepted criteria
* Clinical stability (absence of exacerbations) for at least 3 months before inclusion in the study
* Absence of orthopedic comorbidities which could interfere on the performance of the proposed assessments

Exclusion Criteria:

* Patients will be excluded of the study if they do not demonstrate physical or cognitive conditions to complete the proposed assessments,
* If they suffer from a moderate or severe acute exacerbation in the period between the two assessment points
* If they decide to leave the study for any reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample will be composed by at least 35 patients with moderate-severe COPD from each institution involved (Catholic University of Leuven, Belgium and State University of Londrina, Brazil), adding up to 70 patients. However, the sample size could be increased if necessary to achieve intermediate calculation of the sample power performed during the study. Both groups should be similar concerning anthropometric characteristics, gender distribution and severity feature of the disease (especially FEV1). Therefore, an eventual increase in the final number of patients may also be necessary in case this similarity is not achieved in the final data collection of the planned sample.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Physical activity in daily life | January 2013 and July 2013. Participants will be followed for the duration of 6 months.
  Two activity monitors (the SenseWear armband and the Fitbit) will be simultaneously worn during 7 consecutive days. The SenseWear armband (BodyMedia, Pittsburg, PA, USA) is a multisensor composed by a biaxial accelerometer and physiologic sensors. It is a small (8.8 x 5.6 x 2 cm) and lightweight (82g) monitor that was already validated for energy expenditure estimation in patients with COPD. The Fitbit (Fitbit, Inc., San Francisco, CA, USA) is a recently released triaxial accelerometer that is smaller (3.6 x 2.9 x 1 cm) and more lightweight (8g) than the SenseWear. This device provides the number of steps, the distance walked and the energy expenditure in calories, among other variables. In the 7 days of assessment, the patient will remain with the device during 24 hours/day. The patients will be strictly instructed to avoid changing their daily physical activity habits during the monitoring period.

SECONDARY OUTCOMES:
Six minute walking test | January 2013 and July 2013. Participants will be followed for the duration of 6 months.
  Two tests will be performed with 30 minutes of interval, according to international standards. Subjects will be encouraged to walk during 6 minutes as fast as possible in a straight leveled 30-meter corridor. Reference values will be those by Troosters et al.
Spirometry | January 2013 and July 2013. Participants will be followed for the duration of 6 months.
  Pulmonary function test (post-bronchodilator spirometry) measuring slow vital capacity (SVC), forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), and FEV1/FVC ratio will be performed by the use of a hand-held spirometer (Spiropalm, Cosmed, Italy), following the American Thoracic Society - European Respiratory Society (ATS-ERS) standardized protocol [14] and based on the reference values by Pereira et al. for Brazilian patients and Knudson et al. for European patients.
Chronic Respiratory Disease Questionnaire (CRQ) | January 2013 and July 2013. Participants will be followed for the duration of 6 months.
  The CRQ contains 20 questions divided in 4 domains: dyspnea (5 questions), fatigue (4 questions), emotional function (7 questions) and self control (4 questions). The dyspnea domain is individualized, which means that each patient selects from a list the activities which induce dyspnea in the last two weeks, and they can report other activities that are not on the list. Subsequently, among the reported and selected activities, the patient chooses 5 activities considered the most important ones and by the use of a scale of 7 points the patient grades how much dyspnea interferes on these activities. In this scale the score ranges from 1 (maximum impairment) to 7 (no impairment at all). Concerning the other domains (fatigue, emotional function and self control), the questions are standardized and the patient answers each question using the scale of 7 points. The results are presented on average score of each domain, and the higher the score, the better the subject quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Pitta, PhD, Study Chair — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Karina C. Furlanetto, PT, Study Director — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Nidia A. Hernandes, PhD, Principal Investigator — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Thais Sant'Anna, MSc, Principal Investigator — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Vanessa S. Probst, PhD, Principal Investigator — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Thierry Troosters, PhD, Study Chair — University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Belgium; Heleen Demeyer, PT, Study Director — University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Belgium; Carlos A. Camillo, MSc, Principal Investigator — University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Belgium; Miek Hornickx, PT, Principal Investigator — University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Belgium
Locations (2):
- University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Belgium, Leuven, Belgium
- University Hospital Londrina , Universidade Estadual de Londrina, Brasil, Londrina, Paraná, Brazil